CLINICAL TRIAL: NCT04834076
Title: Genetic Diversity of Toxoplasma Gondii in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Fathi Fadel Mohammed, Teaching assistant of medical parasitology, Sohag University
Other Study IDs: Toxoplasma gondii genomics
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Toxoplasma Gondii Infection; Cancer
MeSH Terms: conditions — Toxoplasmosis; Neoplasms | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples in EDTA tubes for molecular detection of Toxoplasma gondii gene then for sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients: 50 cancer patients referred to the Oncology Department, Faculty of medicine, Sohag University.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: PCR; Diagnostic Test: Sequencing
- Healthy controls: 50 healthy controls will be recruited in the study.
  Interventions: Diagnostic Test: ELISA; Diagnostic Test: PCR; Diagnostic Test: Sequencing

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA is is a test that detects and measures toxoplasma IgG and IgM antibodies in blood.
Diagnostic Test: PCR — Polymerase chain reaction (PCR) is a method widely used to rapidly make millions to billions of copies of a specific DNA sample, allowing scientists to take a very small sample of DNA and amplify it to a large enough amount to study in detail.
Diagnostic Test: Sequencing — DNA sequencing is a laboratory technique used to determine the exact sequence of bases (A, C, G, and T) in a DNA molecule. The DNA base sequence carries the information a cell needs to assemble protein and RNA molecules. DNA sequence information is important to scientists investigating the functions of genes.

SUMMARY:
I. Evaluation of T. gondii infection in cancer patients using different serological markers.

II. Studying genetic lineages infecting cancer patients in Sohag Governorate to predict clinical course and therapeutic needs using B1 and RE genes.

DETAILED DESCRIPTION:
The global cancer burden is estimated to have risen to 18.1 million new cases and 9.6 million deaths in 2018. Patients with cancer have deficient cellular immunity and are potentially susceptible to opportunistic infections including Toxoplasma gondii (T. gondii). Few reports are available about toxoplasmosis in this group of patients. In recent years, it has emerged as an important life-threatening opportunistic pathogen in immunocompromised patients.

T. gondii is a ubiquitous obligate intracellular protozoan parasite that can infect virtually any nucleated vertebrate cell. T. gondii is one of the most successful parasites worldwide, with upwards of 30% of the human population infected.

While T. gondii infection in immunocompetent individuals is usually asymptomatic, it is more detrimental in immunocompromised individuals, such as those with HIV, patients receiving organ transplants or undergoing cancer treatment. A variety of malignancies, including lymphoma, leukemia, and myeloma, can reactivate toxoplasmosis. Moreover, T. gondii is incriminated to be responsible for the progression of malignant diseases.

Screening of toxoplasmosis in cancer patients is mandatory to guard against life-threatening disseminated disease. Diagnosis rely mainly on serology. A study in 2018 was performed to assess the prevalence of anti-T. gondii antibody among cancer patients in Cairo-Egypt. Among 180 cancer patients, a total of 110 patients (61.1%) were positive for anti-T. gondii antibodies. Till now there is no screening program in Egypt for toxoplasmosis in cancer patients although recently demonstrated to be at high risk for acquiring the infection with life-threatening sequelae.

Despite the significant improvements in serological methods, there are still unresolvable limitations such as inability of these methods to confirm the presence of parasite in immunocompromised patients. To overcome these limitations, different molecular methods including conventional PCR (cn PCR), nested PCR, real-time PCR (qPCR) and also loop-mediated isothermal amplification (LAMP) techniques have been developed to detect T. gondii DNA in biological samples.

As molecular diagnosis is not depending on the immunological condition of the host, it would be ideal for cancer patients. The ability of molecular methods to detect low amounts of parasites in fluids or tissues is a key issue, as Toxoplasma can circulate at low concentrations, or inconstantly.

T. gondii has been considered a single species in the genus Toxoplasma. Early studies on the parasite strains from North America and Europe identified limited genetic diversity, which were classified into three clonal lineages I, II, and III.

Genotyping of isolates from all continents revealed a complex population structure. Recent research supports the notion that T. gondii genotype may be associated with disease severity. The outcome of toxoplasmosis is related primarily to host and parasite genetics.

The first PCR technique for T. gondii detection was established by Burg and colleagues in which the 35-repeat B1 gene of T. gondii genome was amplified. Following it, several multi-copy targeting genes including 18S rRNA-, P30-,529-bp repeat fragment or the AF146527 element have been used for the detection of T. gondii in different biological samples.

In spite of the growing data concerning T. gondii genotypes and its role in epidemiological and biological studies,very few studies have been reported in Egypt until now. It is essential to genetically define and characterize T. gondii strains isolated from cancer patients to understand the population genetic structure, population biology, and pathogenesis of this important pathogen in our locality using the highly sensitive molecular techniques.

To the best of our knowledge, this is the first study in Egypt to reveal the population structure of T. gondii in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic cancers on treatment
* Solid Cancers on treatment

Exclusion Criteria:

* Patients with other immune compromise states eg. DM, autoimmune diseases
* Patients who are HIV positive

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 cancer patients referred to the Oncology Department, Faculty of medicine, Sohag University and 20 healthy controls will be recruited in the study.
  Relevant demographic and clinical data will be obtained from all participants. Written consents will be obtained from each participant after clear full explanation about the procedures and their significance.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Isolation and genotyping of T. gondii from blood of Cancer patients in Sohag Governorate, Egypt using PCR and DNA sequencing of Toxoplasma gondii B1 & RE genes. | up to 1 year
  Using PCR and DNA sequencing
Evaluation of T. gondii infection in cancer patients using ELISA. | up to 1 year
  IgG, IgM.

CONTACTS AND LOCATIONS:
Overall Officials: Eman FF Mohammed, Ass lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospitals, Sohag, Egypt